CLINICAL TRIAL: NCT00921921
Title: Does Extra-fine HFA-BDP Suppress Small Airways Inflammation in COPD?
Brief Title: Does Extra-fine Hydrofluoroalkane-beclomethasone Dipropionate (HFA-BDP) Suppress Small Airways Inflammation in Chronic Obstructive Pulmonary Disease (COPD)?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PAW002
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extra-fine particle steroid inhaler (Experimental)
  Interventions: Drug: HFA-BDP
- Placebo control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HFA-BDP — HFA-BDP 100 mcg bid for 3 weeks, then 400 mcg bid for 3 weeks
  Other Names: Qvar
  Arms: Extra-fine particle steroid inhaler
Drug: Placebo — 1 puff bid for 3 weeks, then 1 puff bid for 3 weeks
  Arms: Placebo control

SUMMARY:
Chronic obstructive pulmonary disease or 'COPD' is a chronic disease, which means that it cannot be cured, but that inhalers and tablets can be used to control the symptoms. In COPD, the airways become inflamed which can cause coughing and make the airways tighten. This 'inflammation' is the root of the problem in COPD.

The airways of the lung start in the windpipe and branch like the branches of a tree, getting smaller and smaller. In COPD the inflammation is deep in the lungs, out to the very small airways.

Different inhalers make the medicines into different sized particles. Most steroid inhalers used for COPD make the medicine into particles which are too big to get into the very small airways ('coarse particles'). Other inhalers make a mist, with much smaller particles ('fine particles'). These are as small as the smallest airways in the lungs.

Doctors have recently found a way to measure the inflammation in the small airways that are affected in COPD. The investigators want to find out if taking one of these 'fine-particle' steroid inhalers can treat that inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Current or ex-smokers
* > 40 years of age with a greater than 15 pack year history of smoking
* post-bronchodilator FEV1/FVC ratio < 0.7
* FEV1 < 80% predicted
* CANO > 3 ppb at screening
* Informed consent and ability to perform exhaled nitric oxide assessment

Exclusion Criteria:

* Oral steroid use or exacerbation within 6 weeks
* Greater than 2 exacerbations requiring treatment in the previous 6 months
* Requirement for domiciliary oxygen
* Pregnancy or lactation
* Known or suspected contra-indication to any of the IMP's
* Diagnosis of asthma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Alveolar Nitric Oxide | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asthma and Allergy Research Group, University of Dundee, Dundee, Tayside, United Kingdom

REFERENCES:
- [Result] Short PM, Williamson PA, Lipworth BJ. Effects of extra-fine inhaled and oral corticosteroids on alveolar nitric oxide in COPD. Lung. 2012 Aug;190(4):395-401. doi: 10.1007/s00408-012-9378-8. Epub 2012 Feb 22. PMID 22350679